CLINICAL TRIAL: NCT05213351
Title: Comparison of the Effectiveness of Two Different Exercise Training in Frozen Shoulder Treatment
Brief Title: Two Different Exercise Training in Frozen Shoulder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Zeynal YASACI, Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16.01.2022
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Adhesive Capsulitis
Keywords: frozen shoulder; exercise; graded motor imagery
MeSH Terms: conditions — Bursitis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Motor İmagery (Experimental): Graded Motor İmagery (GMI) group will receive a treatment protocol consisting of Graded Motor Imagery, cold therapy, traditional exercises and home exercises.
  Interventions: Other: Graded Motor Imagery
- Exercise (Active Comparator): Exercise group will receive training involves mobilizations, stretching, specific exercises for the frozen shoulder.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Graded Motor Imagery — Graded Motor Imagery program will be performed two times a week for six consecutive weeks and will include the following three steps: laterality training, imagined movements, and mirror therapy.
  1. Right-left discrimination training (lateralization training)
  2. Imagination of hand movements (motor imagery):
  3. Mirror therapy Treatments including traditional physiotherapy approaches; joint mobilizations, stretching, scapula focused exercises etc.
  Arms: Graded Motor İmagery
Other: Exercise — Treatments including traditional physiotherapy approaches; joint mobilizations, stretching, scapula focused exercises etc.
  Arms: Exercise

SUMMARY:
The aim of this study is to compare the effects of two different exercise programs in patients with frozen shoulders.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed and meet the inclusion criteria will be randomized a double-blind manner in a 1:1 (participant and investigator) to graded motor imagery or exercise group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >60 years
* Patients with shoulder pain of at least six months' duration secondary to tendinopathy and/or partial rotator cuff tear;
* Patients with ability to follow simple orders; iii)
* Patients with ability to sign to provide informed consent

Exclusion Criteria:

* Normal passive ROM
* External ROM < 30
* To have received treatment (physiotherapy, intra-articular injection, surgery) related to the existing complaint
* Pain < 3 according to the numbered pain assessment scale

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline The Shoulder Pain and Disability Index at 6th and 8th week | Baseline,6th week and 8th week
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.

SECONDARY OUTCOMES:
Change from baseline NPRS at 6th and 8th week | Baseline,6th week and 8th week
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.
Change from baseline range of motion at 6th and 8th week | Baseline,6th week and 8th week
  Range of motion is the capability of a joint to go through its complete spectrum of movements.
Change from baseline QuickDASH at 6th and 8th week | Baseline,6th week and 8th week
  The purpose of the QuickDASH is to use 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.
Change from baseline two-point discrimination at 6th and 8th week | Baseline,6th week and 8th week
  The two-point discrimination test is used to assess if the patient is able to identify two close points on a small area of skin, and how fine the ability to discriminate this are. It is a measure of tactile agnosia, or the inability to recognize these two points despite intact cutaneous sensation and proprioception.
Change from Pain Catastrophizing Scale at 6th and 8th week | Baseline,6th week and 8th week
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain.
Change from SF-12 at 6th and 8th week | Baseline,6th week and 8th week
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Çelik, Study Director — Istanbul University
Locations (1):
- İstanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Yasaci Z, Celik D. Does Integration of Graded Motor Imagery Training Augment the Efficacy of a Multimodal Physiotherapy Program for Patients With Frozen Shoulder? A Randomized Controlled Trial. Clin Orthop Relat Res. 2025 Apr 1;483(4):707-716. doi: 10.1097/CORR.0000000000003252. Epub 2024 Sep 17. PMID 39436270